CLINICAL TRIAL: NCT00004166
Title: Amifostine as a Toxicity Protectant in Ovarian Cancer in Chemotherapy Treated Patients: A Pilot Phase III Randomized Controlled Trial
Brief Title: Amifostine in Treating Patients With Ovarian Epithelial Cancer Who Are Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: NU 97CC4; NU-97CC4; NCI-G99-1633
Record Dates: First submitted 1999-12-10; First posted 2004-04-12 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Ovarian Cancer; Quality of Life
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; quality of life
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: amifostine trihydrate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Randomized phase III trial to study the effectiveness of amifostine in treating patients who have ovarian epithelial cancer and who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if patients with ovarian epithelial cancer receiving chemotherapy have significantly fewer neurologic events when treated with amifostine. II. Compare amifostine vs no chemoprotection in terms of overall incidence of neuropathy, incidence of neutropenia, infection, and other myelosuppressive events (e.g., leukopenia, anemia, and thrombocytopenia), length of hospital stay due to infections, and quality of life in this patient population.

OUTLINE: This is a randomized, parallel, controlled, double blind study. Patients are randomized to one of two treatment arms. Arm I: Patients receive amifostine IV over 10 minutes, 30 minutes prior to chemotherapy. Arm II: Patients receive a placebo IV over 10 minutes, 30 minutes prior to chemotherapy. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed prior to courses 1, 4, and 8, and then every 3 months for 1 year. Patients are followed monthly for 6 months.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, surgically staged ovarian epithelial cancer Planned treatment with paclitaxel/carboplatinum chemotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 3 mg/dL SGOT/SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics Other: At least 24 hours since prior antihypertensives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Fishman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States